CLINICAL TRIAL: NCT00020761
Title: A Phase II Study Of Irinotecan (Camptosar) And Paclitaxel (Taxol) In Patients With Adenocarcinoma Of The Upper Gastrointestinal Tract
Brief Title: Irinotecan and Paclitaxel in Treating Patients With Metastatic or Recurrent Cancer of the Esophagus or Stomach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Randolph Hecht, MD / Principal Investigator, UCLA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068711; UCLA-0001048; NCI-G01-1957
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Irinotecan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gastro Esophogeal cohort (Experimental): Patients with adenocarcinoma of the esophagus, gastroesophageal (GE) junction and gastric cardia (GE cohort)
  The course length is 3 weeks. Treatment will continue until one or more of criteria listed in the protocol are met.
  Irinotecan 225 mg/m2 will be infused over 90 minutes every three weeks.
  Paclitaxel 100 mg/m2 will be infused over three hours following irinotecan infusion every three weeks.
  Interventions: Drug: irinotecan hydrochloride; Drug: paclitaxel
- Distal Stomach cohort (Experimental): Patients with adenocarcinoma of the rest of the stomach (Distal Stomach cohort)
  The course length is 3 weeks. Treatment will continue until one or more of criteria listed in the protocol are met.
  Irinotecan 225 mg/m2 will be infused over 90 minutes every three weeks.
  Paclitaxel 100 mg/m2 will be infused over three hours following irinotecan infusion every three weeks.
  Interventions: Drug: irinotecan hydrochloride; Drug: paclitaxel

INTERVENTIONS:
Drug: irinotecan hydrochloride — The course length is 3 weeks. Treatment will continue until one or more of criteria listed in the protocol are met.
  Irinotecan 225 mg/m2 will be infused over 90 minutes every three weeks.
Drug: paclitaxel — The course length is 3 weeks. Treatment will continue until one or more of criteria listed in the protocol are met.
  Paclitaxel 100 mg/m2 will be infused over three hours following irinotecan infusion every three weeks.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining irinotecan and paclitaxel in treating patients who have metastatic or recurrent cancer of the esophagus or stomach.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of irinotecan and paclitaxel in patients with metastatic or recurrent adenocarcinoma of the esophagus or stomach.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to diagnosis (adenocarcinoma of the esophagus, gastroesophageal junction, or gastric cardia vs adenocarcinoma of the rest of the stomach).

Patients receive irinotecan IV over 90 minutes followed by paclitaxel IV over 3 hours on day 1. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 26-54 patients (13-27 per stratum) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Patients with histologic proof of adenocarcinoma of the esophagus (including GE junction) or adenocarcinoma of the stomach will be eligible.
* Location of the tumor for assignment to study will be determined by prior endoscopy or barium contrast study.
* Patients must have either metastatic or recurrent cancer.
* Patients must have bidimensionally measurable disease, as defined in Section 8.4.1.1, page 16. Mediastinal or hilar lymph nodes assessed by CT or MRI scans must be at least 2 cm in the largest dimension to be considered measurable.
* Prior limited radiation therapy is permitted. Prior radiotherapy must not have included major bone marrow containing areas (pelvis, lumbar spine), or contained the single evaluable lesion in a radiation field. A recovery period of at least 4 weeks after completion of radiotherapy is required prior to study treatment.
* Patients must have an anticipated life expectancy of at least 12 weeks.
* Patients must have a performance status of 0 or 1 on the ECOG performance scale.
* Patients must be > 18 years old.
* Patients must give written informed consent prior to enrollment.
* Patients should have adequate organ function defined as follows: Absolute granulocytes > 1,500/mm3 and platelets > 100,000/mm3; serum bilirubin < 1.5 mg/dL and SGOT < 3X upper limit of institutional norm; and serum creatinine < 1.5 mg/dL.
* Patients must have recovered from recent surgery. One week must have elapsed from the time of a minor surgery and 3 weeks from major surgery.

Exclusion Criteria

* Patients who have received more than one prior chemotherapy regimen or immunotherapy for metastatic disease. Prior 5-FU alone as an adjuvant therapy or radiosensitizer is not counted. Patients must have an interval of 4 weeks from prior chemotherapy or immunotherapy with full recovery.
* Patients receiving concurrent chemotherapy, immunotherapy, or radiotherapy.
* Patients who are potentially curable with a chemotherapy, radiotherapy, surgery, or any combination of the above.
* Patients with known brain metastases.
* Patients with a history of seizures or are receiving phenytoin, phenobarbital, or other antiepileptic prophylaxis.
* Pregnant or lactating women. All women of childbearing potential must have a negative pregnancy test prior to entry into the study. All patients of procreative potential must be advised of the importance of avoiding pregnancy and using appropriate methods of contraception while participating in this investigational trial.
* Patients with serious intercurrent infections, or any other concurrent disease which, in the investigator's judgment, would make the patient inappropriate for entry into this study.
* Patients with psychiatric disorders rendering them incapable of complying with the requirements of the protocol.
* Patients with osseous metastasis as only site of disease.
* Patients with any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial.
* Patients with known Gilbert's syndrome.
* Patients who have a significant clinical neuropathy of greater than grade 2.
* Patients with unstable angina, a history of myocardial infarction within the previous 6 months, or current clinical evidence of congestive heart failure. Patients taking medication for congestive heart failure and showing no clinical signs or symptoms are eligible.
* Patients who have previously received a taxane or campthothecin
* Patients who have received any investigational therapy within the previous 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2000-04; Primary Completion 2002-12 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
To determine the antitumor activity of irinotecan and paclitaxel in patients with unresectable adenocarcinoma of the esophagus and gastric cardia. | 5 months

SECONDARY OUTCOMES:
To evaluate the toxicities of irinotecan and paclitaxel in this patient population. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel R. Hecht, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (4):
- United States (4):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - OHSU Cancer Institute, Portland, Oregon